CLINICAL TRIAL: NCT03205306
Title: Myasthenia Gravis and Psyche
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: NeuroCure Clinical Research Center, Charite, Berlin (Other)
Responsible Party: Principal Investigator, Andreas Meisel, Prof. Dr. med., Charite University, Berlin, Germany
Other Study IDs: PsyMG
Record Dates: First submitted 2017-06-08; First posted 2017-07-02 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Myasthenia Gravis
Keywords: Myasthenia Gravis; Psyche; Depression; Anxiety Disorder; Posttraumatic Stress Disorder; Disease Processing
MeSH Terms: conditions — Myasthenia Gravis; Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to systematically capture and characterize mental comorbidities for patients with myasthenia gravis. Anxiety disorders and depression for example, can negatively affect the quality of life and lead to e.g. unemployment and early retirement especially in young patients.

Additionally the researchers want to find out in what way certain aspects of the disease have an influence on the quality of life, and whether different concepts of coping with the disease have different effects on the quality of life for patients with myasthenia gravis.

During the study, close relatives of patients will also be asked to provide input about their current stress situation in the context of supporting their relative.

Based on the results, the investigators want to improve and supplement established treatment concepts, to ensure a more comprehensive and individual treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Myasthenia Gravis
* Age ≥18 years

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Myasthenia Gravis and their relatives
Sampling Method: Probability Sample
Enrollment: 1399 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2017-12-14 (Actual); Study Completion 2017-12-14 (Actual)

PRIMARY OUTCOMES:
Questionnaire Survey (Patient) | directly after inclusion in the study
  * Questionnaire for self-completion by patients containing questions about general information, information on myasthenia, information on diagnosis of mental illness and psychotherapeutic care
  * Hospital Anxiety and Depression Scale (HADS - questionnaire for self-completion by patients to determine the levels of anxiety and depression)
  * Breslau scale PTBS-7 (questionnaire for self-completion by patients to determine the levels of Probability of posttraumatic stress disorder (PTSD))
  * Mya Quality of Life 15 (Mya QoL15 - questionnaire for self-completion by patients for use as a measure of health outcome)
  * Freiburg questionnaire for coping (FKV - questionnaire is used to assess disease processing modes at the levels of cognition, emotion, and behavior)

SECONDARY OUTCOMES:
"Häusliche Pflegeskala" (HPS) | directly after inclusion in the study
  questionnaire is used to assess social work Intervention and couple's counselling

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Meisel, Prof. Dr. med., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- NeuroCure Clinical Research Center (NCRC), Charité, Berlin, Germany

REFERENCES:
- [Result] Marbin D, Piper SK, Lehnerer S, Harms U, Meisel A. Mental health in myasthenia gravis patients and its impact on caregiver burden. Sci Rep. 2022 Nov 11;12(1):19275. doi: 10.1038/s41598-022-22078-3. PMID 36369246